CLINICAL TRIAL: NCT01723709
Title: The MURDOCK Study Community Registry and Biorepository Multiple Sclerosis Cohort
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00023791
Record Dates: First submitted 2012-10-24; First posted 2012-11-08 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-06

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; immune response; genetic; progression; relapse; biomarkers; disease; proteomics; genome; gene
MeSH Terms: conditions — Multiple Sclerosis; Disease Progression; Recurrence; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 7.5 mL PaxGene RNA collection 6 mL DNA whole blood collection 40 mL urine collection 20 mL serum SST tube collection 16 mL plasma EDTA tube collection
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this study is to enroll 1000 participants with a history of Multiple Sclerosis into the MURDOCK Study (Duke IRB Pro00011196) as well as into the Multiple Sclerosis Cohort study (Duke IRB Pro00023791). All 1000 participants will answer a 4-page questionnaire administered by a trained study coordinator which is designed to collect information on the participant's diagnosis of Multiple Sclerosis. The goal of the study is to seek genetic explanations for response to treatment, progression of the disease, and biomarker validation.

DETAILED DESCRIPTION:
Despite tremendous research efforts, the targets of immune response and the mechanisms for neuronal loss associated with MS have not been fully characterized. Although substantial advances have been made in the development of therapeutic treatments, the drugs currently available to MS patients do not significantly alter the long-term prognosis of the disease. Better markers that represent the biological activity of the disease process and response to therapy are desperately needed. MS is thought to be mediated by autoimmunity which causes demyelination and transection of axons throughout the brain and spinal cord resulting in the formation of multiple scars (or scleroses) on axon myelin sheaths and reducing electrical conductivity and decreased CNS signaling. It is most common in young adults; more than 90% of patients are diagnosed before the age of 55 and less than 5% before the age of 14. Females are 2-3 times more frequently affected than males and children of affected females are at a significantly higher risk of developing MS than children of affected males. A strong genetic component is suggested by the co-occurrence of cases within families and the high disease prevalence in some ethnic populations (particularly those of northern European origin) compared with others (African and Asian groups) irrespective of geographic location.7 The incidence of MS in northern Europe, where the genetically associated haplotype HLA DR2 is most common, is as high as 1 per 750 individuals. MS affects more than 400,000 people in the U.S. and 2.5 million worldwide.

Although numerous putative MS-specific biomarkers, representing different mechanisms of pathogenesis and steps along the inflammatory cascade have been proposed, none have been fully validated. To date, the majority of studies identifying biomarkers associated with MS initiation or progression have been limited to investigation of one to several markers at a time; only one study has attempted open platform proteomic profiling in MS; however, the study size was relatively small and the clinical homogeneity of the dataset of the study is not clear. To understand a complex disease like MS, high throughput technologies capable of profiling multiple etiological changes is needed as well as a well-define population of those with the disease.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Multiple Sclerosis Diagnosis or self report Multiple Sclerosis

Exclusion Criteria:

* Participants who are not willing to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants must enroll or have enrolled in the MURDOCK Study Community Registry and Biorepository prior to joining the Multiple Sclerosis Cohort. At the MURDOCK Study visit, or after the participant has enrolled in the MURDOCK Study, they will be asked (either in person or via the phone) if they would be willing to join the Multiple Sclerosis cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 973 (Actual)
Dates: Start 2010-06; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Serum-based proteomic biomarkers associated with disease initiation and progression in MS | 5 years
  Biological material (serum, urine, whole blood and Paxgene RNA) collected in the MURDOCK Study(Pro00011196) will permit the initiation of a biomarker discovery project for all patients consented under the MS cohort protocol. Participants in this study will be followed for 5 years after consent with additional blood draws and questionnaires occurring biannually during this period.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Gregory, PhD, Principal Investigator — Duke Medicine Site Based Research Group
Locations (5):
- United States (5):
  - Carolinas Medical Center Northeast Medical Arts Building, Concord, North Carolina
  - Ada Jenkins Center, Davidson, North Carolina
  - The Stedman Center on the Duke Center for Living Campus, Durham, North Carolina
  - Kannapolis Internal Medicine, Kannapolis, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina